CLINICAL TRIAL: NCT04205669
Title: A Randomized Controlled Trial Comparing the Effectiveness of Individual vs. Household Treatment for Scabies in Lambaréné, Gabon
Brief Title: Comparing the Effectiveness of Individual vs. Household Treatment for Scabies in Lambaréné, Gabon
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Collaborators: Bernhard Nocht Institute for Tropical Medicine (Other Government); University Hospital Tuebingen (Other); Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Julian Matthewman, Principal Investigator, Centre de Recherche Médicale de Lambaréné
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GrattiGratta31082018
Record Dates: First submitted 2019-12-18; First posted 2019-12-19 (Actual); Results first posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Scabies; Households
MeSH Terms: conditions — Scabies | interventions — benzyl benzoate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individual Treatment (Active Comparator)
  Interventions: Drug: Benzyl Benzoate 25% Topical Application Lotion
- Household Treatment (Active Comparator)
  Interventions: Drug: Benzyl Benzoate 25% Topical Application Lotion

INTERVENTIONS:
Drug: Benzyl Benzoate 25% Topical Application Lotion — Applied to skin for the treatment of scabies

SUMMARY:
It is unclear whether individual treatment of scabies is similarly effective compared to household treatment. This study therefore compares these two treatment strategies with topical benzyl benzoate for treating scabies in Lambaréné and surroundings in Gabon.

Subjects presenting with uncomplicated scabies are randomized into either the Individual Treatment group, where only the affected subjects receive treatment, or the Household Treatment group, where all family members are treated in parallel to the affected subjects regardless of signs and symptoms. The primary endpoint is clinical cure after 28 days; the secondary endpoint is the proportion of affected household members per household after 28 days.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with active, uncomplicated scabies
* no known hypersensitivity or allergy against benzyl benzoate

Exclusion Criteria:

* hypersensitivity or allergy against benzyl benzoate
* severe superinfection of scabies lesions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherches Médicales de Lambaréné, Lambaréné, Gabon

IPD SHARING:
Plan to Share IPD: Yes
IPD with identifying data removed uploaded to public repository under https://www.kaggle.com/julianmatthewman/grattigratta-data
URL: https://www.kaggle.com/julianmatthewman/grattigratta-data

REFERENCES:
- [Derived] Matthewman J, Manego RZ, Dimessa Mbadinga LB, Sinkovec H, Volker K, Akinosho M, Haedrich C, Tardif d'Hamonville J, Lell B, Adegnika AA, Ramharter M, Mombo-Ngoma G. A randomized controlled trial comparing the effectiveness of individual versus household treatment for Scabies in Lambarene, Gabon. PLoS Negl Trop Dis. 2020 Jun 26;14(6):e0008423. doi: 10.1371/journal.pntd.0008423. eCollection 2020 Jun. PMID 32589632
- Available data/document: Individual Participant Data Set — https://www.kaggle.com/julianmatthewman/grattigratta-data

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individual Treatment | Household Treatment
Started | 47 | 57
Completed | 34 | 45
Not Completed | 13 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individual Treatment | Household Treatment | Total
Number analyzed (Participants) | 47 | 57 | 104
Age, Customized [Count of Participants; unit: Participants]
  <12 years | 29 | 36 | 65
  >=12 years | 18 | 21 | 39
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 30 | 52
  Male | 25 | 27 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Scabies severity [Count of Participants; unit: Participants]
  Mild | 6 | 5 | 11
  Moderate | 19 | 31 | 50
  Severe | 22 | 21 | 43
Malaria rapid diagnostic test status [Count of Participants; unit: Participants]
  Positive | 22 | 16 | 38
  Negative | 25 | 41 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Cure
Description: clinical improvement in skin lesions with no new lesions occurring since treatment application as assessed by skin examination
Time Frame: after 28 days from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Individual Treatment | Household Treatment
Number analyzed (Participants) | 34 | 45
Participants | 20 | 33

2. Secondary Outcome: Proportion of Affected Household Members Per Household
Description: proportion of scabies cases per household after 4 weeks
Time Frame: after 28 days from baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: over the study follow up period, an average of 4 weeks
Arm/Group | Individual Treatment | Household Treatment
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/57
Other Adverse Events (participants affected / at risk) | 0/47 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/69/NCT04205669/Prot_SAP_000.pdf